CLINICAL TRIAL: NCT01906840
Title: Evaluate the Effects of Turmeric on Oxidative Stress Markers in HD Patients
Brief Title: Role of Turmeric on Oxidative Modulation in ESRD Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Maryam Pakfetrat, associated professor of shiraz Shiraz University of Medical Sciences, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Interventional; 2483 (Other: snurc)
Record Dates: First submitted 2013-07-21; First posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: End Stage Renal Failure
Keywords: Chronic renal failure; Hemodialysis; Oxidative stress; Turmeric
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- drug: turmeric capsule (Experimental): Intervention is turmeric (one capsule with each meal containing 500 mg turmeric, of which 22.1 mg was the active ingredient curcumin; three capsules daily) for 8 weeks
  Interventions: Drug: Turmeric
- Drug: placebo,capsule (Placebo Comparator): Intervention is daily starch capsules 500 mg for 8 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Turmeric
  Arms: drug: turmeric capsule
Drug: placebo
  Arms: Drug: placebo,capsule

SUMMARY:
Despite advances in prevention of cardiovascular diseases, the incidence of accelerated atherosclerosis in hemodialysis (HD) patients has still remained high. Oxidative stress is considered as a major player in uremia associated morbidity and mortality in HD patients. The aim of this study was to evaluate the effects of turmeric on oxidative stress markers in HD patients.

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) is a state of oxidative stress, due to uremic oxidant mediator's accumulation, the activation of phagocytic oxidative metabolism by the dialysis membrane, intravenous iron therapy and the antioxidant depletion caused by hemodialysis (HD). Some trials showed a significant benefit from antioxidant therapy on cardiovascular outcome in HD patients.

Extensive research focused on direct exogenous antioxidants including vitamin C, and vitamin E, in the treatment of cardiovascular disease. Some clinical trials showed no more beneficial effect of exogenous antioxidant supplementation in cardiovascular disease (CVD) and recommended the necessity for a new approach to regulating cellular redox status.

Turmeric (Curcuma longa Linn) is an herb used as a dietary spice and in traditional medicine for centuries. Curcumin, the most active and non-toxic component of turmeric, is a polyphenol, which has been extensively studied for its therapeutic benefits, such as antioxidant. Besides, turmeric has also been effective in attenuation of proteinurea in diabetic nephropathy and lupus nephritis patients.

Curcumin restored the activities of mitochondrial enzymes complexes and thereby attenuated the release of reactive oxygen species. Turmeric appears to be non-toxic to humans even at high doses. However, there is a paucity of information on the effect of turmeric in HD population. We have, therefore, followed up this study to determine the beneficial effect of turmeric on oxidative stress in HD patients.

ELIGIBILITY:
Inclusion Criteria:

* having the age of 18 years and more,
* receiving 4-hour HD treatments 3 times per week at least for three months,
* administering no other antioxidant medications

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
effects of turmeric on oxidative stress markers | 8 weeks